CLINICAL TRIAL: NCT00294294
Title: A Randomized Controlled Open-Label Phase IV Multi Center Study to Assess the Effect of Antipyretic Prophylactic Treatment on the Rate of Febrile Reactions Following Concomitant Contralateral Administration of a 7-Valent Pneumococcal Conjugate Vaccine (Prevenar®) and DTPa-HBV-IPV+Hib Vaccine (Infanrix Hexa®) in Children at 2, 3, 4 and 11-14 Months of Age
Brief Title: Study Evaluating Treatment of Fever in Children Who Have Been Vaccinated With Prevenar and Infanrix Hexa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6106A1-500
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Vaccines, Pneumococcal; Infant; Fever, Chemically Induced; Drug Therapy, Combination
Keywords: vaccine; infant
MeSH Terms: conditions — Fever | interventions — Heptavalent Pneumococcal Conjugate Vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

INTERVENTIONS:
Biological: Prevenar
Biological: Infanrix hexa

SUMMARY:
The purpose of the study is to determine whether prophylactic antipyretic treatment after vaccination with Prevenar and a concomitant hexavalent DTPa combination vaccine reduces the rate of febrile reactions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants age 55 to 112 days
* Subject's parents/legal guardians provide written informed consent

Exclusion Criteria:

* Prematurely born subjects < 37 weeks gestation
* Known or suspected disease of immune system
* Known or suspected hypersensitivity to any vaccine or vaccine component

Ages: 56 Days to 112 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Start 2005-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Rectal temperature >= 38°C within days 1-4 post vaccination after any of the doses 1-4

SECONDARY OUTCOMES:
Rectal temperature > 39.0°C occurring within 4 days of vaccine administration after each of the doses 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Rose MA, Juergens C, Schmoele-Thoma B, Gruber WC, Baker S, Zielen S. An open-label randomized clinical trial of prophylactic paracetamol coadministered with 7-valent pneumococcal conjugate vaccine and hexavalent diphtheria toxoid, tetanus toxoid, 3-component acellular pertussis, hepatitis B, inactivated poliovirus, and Haemophilus influenzae type b vaccine. BMC Pediatr. 2013 Jun 21;13:98. doi: 10.1186/1471-2431-13-98. PMID 23786774